CLINICAL TRIAL: NCT01473173
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Dose Escalation Study, to Investigate the Safety, Tolerability, PK and PD of Escalating Single and Multiple Oral Doses of CJ-12420 in Healthy Male Subjects
Brief Title: Safety, Tolerability, PK, PD of Escalating Single and Multiple Oral Doses of CJ-12420 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CJ_APA_101
Record Dates: First submitted 2011-11-14; First posted 2011-11-17 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Healthy
Keywords: Safety; Tolerability; Pharmacokinetics; Pharmacodynamics
MeSH Terms: interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- CJ-12420 50mg (Experimental): * Single dose
  * 8 volunteers will be administered CJ-12420 50mg or placebo comparators.(CJ-12420:placebo=6:2)
  Interventions: Drug: CJ-12420
- CJ-12420 100mg (Experimental): * Single dose
  * 8 volunteers will be administered CJ-12420 100mg or placebo comparators.(CJ-12420:placebo=6:2)
  Interventions: Drug: CJ-12420
- CJ-12420 200mg (Experimental): * Single dose
  * 8 volunteers will be administered CJ-12420 200mg or placebo comparators.(CJ-12420:placebo=6:2)
  Interventions: Drug: CJ-12420
- CJ-12420 400mg (Experimental): * Single dose
  * 8 volunteers will be administered CJ-12420 400mg or placebo comparators.(CJ-12420:placebo=6:2)
  Interventions: Drug: CJ-12420
- CJ-12420 100mg (repeated dose) (Experimental): Repeat doses
  * 100mg is the anticipated dose
  * 8 volunteers will be administered CJ-12420 100mg or placebo comparator.(CJ-12420:placebo=6:2)
  Interventions: Drug: CJ-12420
- CJ-12420 200mg (repeated dose) (Experimental): Repeat doses
  * 200mg is the anticipated dose
  * 8 volunteers will be administered CJ-12420 200mg or placebo comparator.(CJ-12420:placebo=6:2)
  Interventions: Drug: CJ-12420
- Esomeprazole 40mg (Active Comparator): 8 volunteers will be administered Esomeprazole 40mg
  Interventions: Drug: Esomeprazole 40mg

INTERVENTIONS:
Drug: CJ-12420
  Arms: CJ-12420 100mg; CJ-12420 100mg (repeated dose); CJ-12420 200mg; CJ-12420 200mg (repeated dose); CJ-12420 400mg; CJ-12420 50mg
Drug: Esomeprazole 40mg
  Other Names: Nexium
  Arms: Esomeprazole 40mg

SUMMARY:
The objectives of this study are:

* To evaluate the safety and tolerability of single and multiple oral doses of CJ-12420 in healthy male subjects.
* To evaluate the single- and multiple-dose PK of orally administered CJ-12420 in healthy male subjects.
* To evaluate the single- and multiple-dose PD of orally administered CJ-12420 in healthy male subjects.
* To compare the multiple-dose pharmacodynamics (PD) of orally administered CJ-12420 and esomeprazole in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male volunteers in the age between 20 and 45 years old (inclusive)
* Body mass index (BMI) in the range of 19 to 28 kg/m2 and weighing at least 50 kg
* Medically healthy with no clinically significant vital signs (sitting position blood pressure, pulse rate) (90 mmHg ≤ systolic blood pressure ≤ 140 mmHg, 50 mmHg ≤ diastolic blood pressure ≤ 95 mmHg, 45 beats per minute ≤ pulse rate ≤ 95 beats per minute)
* Non-smokers or non-users of nicotine-containing products for at least 3 months

Exclusion Criteria:

* History of clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, psychiatric, musculoskeletal or cardiovascular disease or any other condition, which, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results
* History of allergy or sensitivity to any drug, including any prior serious adverse reaction to PPIs (e.g. omeprazole, rabeprazole, lansoprazole)
* History of symptomatic GERD, erosive esophagitis, duodenal ulcer, gastric ulcer, Barrett's esophagus or Zollinger-Ellison syndrome, previous positive H. pylori

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2011-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the PK, PD, safety and tolerability of escalating single and multiple oral doses of CJ-12420 in healthy male subjects | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Kyun-Seop Bae, MD, Ph.D, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea